CLINICAL TRIAL: NCT01580527
Title: A Prospective, Multicentric, Randomized Trial Comparing Early Enteral Nutrition Versus Parenteral Nutrition After Pancreaticoduodenectomy
Brief Title: Postoperative Artificial Nutrition After Pancreaticoduodenectomy
Acronym: Nutri-DPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010.627
Record Dates: First submitted 2012-01-31; First posted 2012-04-19 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Disease
Keywords: postoperative artificial nutrition; parenteral nutrition; enteral nutrition; postoperative complications; cephalic pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Diseases; Hyperphagia; Postoperative Complications | interventions — Parenteral Nutrition, Total; Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- total parenteral nutrition (Active Comparator)
  Interventions: Procedure: Total parenteral nutrition
- Early enteral nutrition (Experimental)
  Interventions: Procedure: Enteral nutrition

INTERVENTIONS:
Procedure: Total parenteral nutrition — Total parenteral nutrition in postoperative of pancreaticoduodenectomy
  Arms: total parenteral nutrition
Procedure: Enteral nutrition — Early enteral nutrition in postoperative of pancreaticoduodenectomy
  Arms: Early enteral nutrition

SUMMARY:
Pancreaticoduodenectomy is a major surgery burdened by important morbidity and mortality partially related to the altered nutritional status of the patients. The perioperative malnutrition is a major risk factor of postoperative complications and worsens the prognosis of the patients. The perioperative artificial nutrition has for objectives to correct the preoperative malnutrition, and to maintain the nutritional status in the post-operative period. The current guidelines in surgery are in favour of a realisation of a perioperative artificial nutrition support that privilege the enteral nutrition. However, after pancreaticoduodenectomy, the total parenteral nutrition remains most usually used in the early postoperative period, although rare studies suggest a benefit of the enteral nutrition in term of reduction of the post-operative complications. Indeed, no recommendation was formulated concerning early enteral nutrition after pancreaticoduodenectomy because few studies were realized on its profits.

The data of the literature report rates of complications (essentially major) from 49 % to 59 % after major digestive surgery (not only pancreatic) on patients having received a total parenteral nutrition versus rates from 34 to 43.8 % in patients having received an early enteral nutrition.

A preliminary prospective study realized in the investigators centre showed a rate of 74 % complication versus 44 %, respectively in the total parenteral nutrition and early enteral nutrition groups (50 patients in every group, with p < 0.01. All the complications were listed prospectively).

Hypothesis :

The early enteral nutrition will allow, after pancreaticoduodenectomy, a decrease of, at least, 19 % complications of any stage according to the classification of Dindo-Clavien (59 % versus 40 %).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients more than 18 years of age.
* Pancreatic surgery by pancreaticoduodenectomy.
* Patient affiliated to a mode of the social security or receiving of such a mode.
* Having given written informed consent prior to any procedure related to the study

Exclusion Criteria:

* ASA score ≥4
* Pregnant women
* Patient who cannot give written informed consent.
* Concomitant participation in a biomedical study being able to interfere with this research
* Patient less than 18 years of age or more than 18 years of age, protected by the Law, under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients presenting one or several postoperative complications | 90 days
  Data recorded during the period of hospitalization (an expected average of 3 weeks) and until control visit 3 months after surgery

SECONDARY OUTCOMES:
Nutritional status | 90 days
  weight, BMI, Index of Nutritional Risk, blood albumin and prealbumin, during the period of hospitalization (an expected average of 3 weeks) and until control visit 3 months after surgery
Infectious complications | within the hospitalization time after surgery (an expected average of 3 weeks)
  Percentage of patients presenting an infectious complication, and type of infectious complication
Evaluation of the severity of the complications | within the hospitalization time after the surgery (an expected average of 3 weeks)
  according to classification of Dindo-Clavien
Pancreatic fistulas | within the hospitalization time after the surgery (an expected average of 3 weeks)
  evaluation of the occurrence of pancreatic fistulas, grade B and C, in both groups of patients
Hemorrhagic complications | within the hospitalization time after the surgery (an expected average of 3 weeks)
  evaluation of the occurrence of hemorrhagic complications, grade B and C, in both groups of patients
gastroparesis | within the hospitalization time after the surgery (an expected average of 3 weeks)
  defined as the presence of the nasogastric probe 10 days after the surgery
Duration of hospital stay | within the hospitalization time after the surgery (an expected average of 3 weeks)
Time frame of resumption of the intestinal bowel motion | within the hospitalization time after the surgery (an expected average of 3 weeks)
  daytime of resumption of flatulencies and\or stools
Time frame of resumption of the oral food and artificial nutrition weaning | within the hospitalization time after the surgery (an expected average of 3 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Unité de Chirurgie Hépatobiliaire et Pancréatique Hopital Edouard Herriot, Lyon, France